CLINICAL TRIAL: NCT03938584
Title: The Effect of Vitamin C on Wound Healing In Mandibular Fracture Patients: A Double Blind, Placebo-controlled Randomized Clinical Trial
Brief Title: The Effect of Vitamin C on Wound Healing In Mandibular Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Regions Hospital (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR# 1-4276
Record Dates: First submitted 2019-04-26; First posted 2019-05-06 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Vitamin C Deficiency; Smoking; Surgery; Surgery--Complications; Wound; Wound Complication; Wound Infection; Wound Dehiscence; Wound of Skin; Mandible Fracture; Mandible Open Fracture; Mandible Closed Fracture; Mandibular Fractures; Ascorbic Acid Deficiency; Oxidative Stress; Inflammation
MeSH Terms: conditions — Ascorbic Acid Deficiency; Smoking; Wounds and Injuries; Wound Infection; Mandibular Fractures; Inflammation | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental)
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Just after induction of anesthesia in the OR, subjects will be administered a single intravenous (IV) dose of Vitamin C at 66mg/kg/hr for 2 hours during surgery. Post-operatively (beginning the morning after surgery) Vitamin C Treatment Group subjects will receive a 4 week prescription of oral, liquid Vitamin C, 500mg by mouth two times a day. These dosages are known to be safe and effective.89-91
  Other Names: Ascorbic Acid
  Arms: Vitamin C
Other: Placebo — Subjects will receive IV placebo (normal saline) identically packaged. Post-operatively Placebo Control Treatment Group participants will receive a 4-week prescription of the aqueous solution base used for the treatment group without the active component (Vitamin C).
  Arms: Placebo

SUMMARY:
The goal of this study is to perform a randomized clinical trial to assess the effects of vitamin C versus placebo on wound healing in mandibular fracture patients.

DETAILED DESCRIPTION:
In a prospective, randomized clinical trial of de novo mandibular fracture patients requiring intraoral surgical repair with plating, the investigators will:

1. Compare the effects of supplemental vitamin C to placebo on soft tissue wound healing, measured by a) biomarkers of soft tissue repair (Procollagen I and III, Matrix Metallo-Proteinases 1,2,3 & 9, C-reactive protein, neutrophil count, Interleukins 6 & 8, TBARS and TEAC) and b) clinical outcomes (wound dehiscence and Wound Score).

   Hypothesis1: Supplemental vitamin C will improve soft tissue healing post-mandibular fracture, measured by improved procollagen I, other biomarker levels and clinical outcomes, compared to placebo.

   Rationale. The clinical literature describes impaired soft tissue wound healing in mandibular fracture patients, including wound infection, wound dehiscence, and plate exposure. Vitamin C is a necessary co-factor for the production of types I and III collagen, as well as procollagen, the precursor to collagen, via the hydroxylation of proline and lysine. In the setting of vitamin C deficiency, collagen production is abnormal leading to defective vessel and connective tissue formation with degradation of unstable collagen molecules.90-91,34, 63, 108,109

   The investigators will collect a robust set of clinical outcomes including clinician evaluation and Wound Healing Score to measure soft tissue healing. Biomarkers of soft tissue wound healing will be used to measure biochemical healing pathways as well. As a precursor to collagen, procollagen I and III are widely used biomarkers of collagen production in wound healing research. The investigators will assess these levels at baseline and at 3 to 5weeks post-operatively to evaluate the effect of vitamin C on collagen production. In addition, the antioxidant effects of vitamin C are critical during the ordered phases of wound healing, from the inflammatory phase (including the initial hemostatic cascade) to the proliferative phase. Antioxidant depletion during these phases results in imbalanced proteolytic enzyme cascades (including matrix metalloproteinases or MMPs) with resulting tissue destruction as well as an over-exuberant inflammatory milieu. Further, the antioxidant deficit resulting from vitamin C deficiency results in diminished monocyte and neutrophil chemotaxis and diminished bacteriocidal oxidative burst capabilities. Thus, the investigators will additionally measure the effects of vitamin C supplementation on proteolytic enzyme pathways (MMPs) and systemic markers of infection and inflammation (neutrophil count, c-reactive protein level, interleukins (IL) 1 and 6). Finally, the investigators will use indicators of oxidative stress at baseline and 6 weeks to measure the effects of vitamin C supplementation on antioxidant capacity (TBARS and TEAC).
2. Compare the effects of supplemental vitamin C to placebo on bone repair, measured by a) biomarkers of bone repair (alkaline phosphatase, TRACP 5b, osteocalcin, RANKL, osteoprotegerin, and carboxy terminal collagen crosslinks) and b) clinical outcomes (radiologic imaging and pain).

   Hypothesis 2: Supplemental vitamin C will improve bone healing post-mandibular fracture, measured by improved biomarkers of bone healing and more robust radiological bone imaging, compared to placebo.

   Rationale. A body of literature, from animal studies to randomized clinical trials, supports the notion that vitamin C is necessary for bone health and healing. Multiple animal studies demonstrate that vitamin C promotes bone formation / mineralization, strengthens developing callous, and supports bone maintenance. Further, a number of studies show that supplemental vitamin C prevents fracture in menopausal women and may be protective against arthritis.10,11,12,69 Several well done randomized controlled clinical trials have shown that supplemental vitamin C diminishes regional pain syndrome after distal radius fractures and less robust data suggests this for foot and ankle fractures. Well-done randomized controlled clinical trials are needed to develop Vitamin C guidelines in traumatic facial fracture.

   The investigators will collect a comprehensive set of biochemical, clinical, and radiological outcome measures to evaluate bony healing after mandibular fracture. The biomarker evaluation will include assessment of osteoblast and osteoclast number (alkaline phosphatase and TRACP 5b respectively), osteoblast activity (osteocalcin), osteoclast differentiation (receptor activator for nuclear factor, B ligand or RANKL and osteoprotegerin or decoy receptor for RANKL) and osteoclast activity (carboxy terminal collagen crosslinks). The investigators will measure clinical outcomes about 1 and 3 to 5 weeks postoperatively. Finally, each subject will undergo a non-contrast CT of the mandible 3to 5 weeks post-operatively for radiological evaluation of bone healing. The CT scan may or may not be standard of care.30,36,135
3. Determine the effects of supplemental vitamin C on soft tissue and bone healing by smoking status in patients with traumatic mandibular fracture.

Hypothesis 3: Current smokers will have a higher prevalence of vitamin C deficiency than nonsmokers at baseline, and vitamin C supplementation will improve soft tissue and bone healing more in smokers than nonsmokers.

Rationale. Despite clinical evidence for smoking-related impairment in wound healing, much is unknown about the pathophysiologic mechanisms underlying this effect.21. It is postulated that after injury, smoking impedes the inflammatory phase of wound healing by diminishing cellular chemotactic responsiveness, migratory function, and oxidative bacterial killing, and by creating an imbalance in protease-protease inhibitor relationships. The proliferative phase of wound healing is also potentially impaired by smoking, with diminished fibroblast proliferation and migration resulting in decreased collagen production.124-30 Increases in oxidative stress and hypoxia further diminish healing in smokers.62,74,76,102 Vitamin C is postulated to be an important contributor to the diminished wound healing evidenced in smokers. Both population and experimental studies have shown smokers are more likely to be deficient in Vitamin C, with 25% of female smokers and 30% of male smokers having severe deficiency. This deficiency is likely secondary to a systemic depletion by the many reactive oxygen species in tobacco smoke as well as a diet lacking antioxidants. The investigators will evaluate the effects of vitamin C on wound healing in current versus non smokers with detailed assessment of tobacco use.

This project assembles a multidisciplinary team with expertise in wound healing, maxillofacial surgery, medical effects of tobacco use, fracture repair, biomechanics of bone, and conduct of clinical trials. The proposed work will define specific effects of supplemental Vitamin C on soft tissue and bone healing, with additional attention to smoking status in patients with mandibular fractures. For the many patients who are at high risk for vitamin C deficiency and poor wound healing, this investigation will provide critical knowledge of the role of oxidative stress and anti-oxidants in the mechanisms of impaired healing. These data will provide pilot data to support randomized controlled trials of interventions to improve post-operative wound healing in patients suffering from mandibular and other traumatic fractures. Establishing the safety and efficacy of supplemental Vitamin C in the peri-operative setting will improve wound healing outcomes for thousands of patients undergoing traumatic fracture surgery and could be a transformative step in treatment guidelines for any smoker undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18 or older with de novo mandibular fracture undergoing surgical repair with an intra-oral incision based approach with plating (ie- not solely mandibular maxillary fixation which requires no surgical incision).,
* surgery within 7 days of injury.

Exclusion Criteria:

* cognitive impairment limiting ability to provide informed consent
* pregnancy or nursing
* a known history of renal insufficiency
* comminuted fractures,
* allergy to Vitamin C / placebo components.
* Isolated subcondylar fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Procollagen I | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in picogram/milliliter (pg/ml) in blood serum.
Procollagen III | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in picogram/milliliter (pg/ml) in blood serum.

SECONDARY OUTCOMES:
Matrix Metallo-Proteinases 1,2,3 & 9 | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in picogram/milliliter (pg/ml) in blood
C-reactive protein | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in nanogram/milliliter (ng/ml) in blood
Neutrophil count | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in picogram/milliliter (pg/ml) in blood
Interleukins 6 & 8 | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in picogram/milliliter (pg/ml) in blood
Thiobarbituric acid reactive substances | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in micro Molar uM in blood
Trolox equivalent antioxidant capacity | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of soft tissue repair. Measured in nanomol/microliter (nmol/ul) in blood
alkaline phosphatase | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of bone repair. Measured in enzyme unit/liter (U/L) in blood
Tartrate Resistant Acid Phosphatase 5b | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of bone repair. Measured in enzyme unit/liter (U/L) in blood
osteocalcin | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of bone repair. Measured in picogram/milliliter (pg/ml) in blood
osteoprotegerin | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of bone repair. Measured in picogram/milliliter (pg/ml) in blood
carboxy terminal collagen crosslinks | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of bone repair. Measured in nanogram/milliliter (ng/ml) in blood
Receptor activator of nuclear factor kappa-B ligand | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of bone repair. Measured in picogram/milliliter (pg/ml) in blood
Vitamin C | Blood is obtained the day of surgery and 6 weeks after surgery
  Vitamin C levels. Measured in nanomols (nmmol) in blood serum
Cotinine | Blood is obtained the day of surgery and 6 weeks after surgery
  Biomarker of tobacco exposure. Measured in nanograms/milliliter (mg/ml) in blood serum.

OTHER OUTCOMES:
Wound score | Wounds are analyzed 1 week and 6 weeks after surgery.
  Wounds are scored from photographs using the InCISE wound score developed by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No